CLINICAL TRIAL: NCT03149432
Title: Effectiveness of Mirror Therapy in Patients With Amputations of Lower Limbs of Vascular Origin
Acronym: MIR-PHAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-A00771-50
Record Dates: First submitted 2017-02-03; First posted 2017-05-11 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-05

CONDITIONS: Amputation; Phantom Pain Following Amputation of Lower Limb
Keywords: mirror therapy; amputation; phantom pain
MeSH Terms: conditions — Phantom Limb | interventions — Mirror Movement Therapy; Gabapentin; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assossor won't know if the participant has received the mirror therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference analgesic (Active Comparator): Gabapentin Rehabilitation Local care
  Interventions: Drug: Gabapentin; Procedure: Rehabilitation; Other: Local care
- reference analgesic and mirror therapy (Experimental): Mirror Therapy Gabapentin Rehabilitation Local care
  Interventions: Procedure: Mirror Therapy; Drug: Gabapentin; Procedure: Rehabilitation; Other: Local care

INTERVENTIONS:
Procedure: Mirror Therapy — by a mirror effect the patient sees his remaining arm at the place of the amputated arm that cause an illusion of presence of this arm to the brain and would have an effect of reducing phantom pain
  Arms: reference analgesic and mirror therapy
Drug: Gabapentin — titration of Gabapentin up to 3600 mg or maximum tolerated dose for 8 weeks
Procedure: Rehabilitation — Daily care with physiotherapist ; orthoprosthetists , and specialized sports educators ; if necessary : occupational therapy.
Other: Local care — local care for directed healing of the stump.

SUMMARY:
The aim of this study is to assess the efficacy of the mirror therapy on phantom pain for patients with amputation after vascular etiology. the secondary aim are to measure the impact of the mirror therapy on quality of life, sleep disorders, and predictive factors for effectiveness. the design is a prospective study, randomised, blindly evaluated, monocentric. There will be 2 groups: 1) rehabilitation and gabapentine; 2) rehabilitation and gabapentine + mirror therapy during the first 4 weeks. The assessment are going to be preformed at the inclusion day and then every 2 weeks during 8 weeks. the primary evaluation criterion will be the phantom pain measured on a VAS. the delay for inclusion is 18 months in order ton include 40 patients. The length of the study is 20 months.

DETAILED DESCRIPTION:
Several variables at the beginning collected to study the predictive factors of effectiveness of mirror therapy:

* Age
* Sex
* Delay from amputation
* Etiology: neuropathy associated or not
* VAS of preoperative pain
* VAS phantom pain at baseline
* Localization of pain
* Ability to mobilize the phantom limb
* Healing obtained or not
* Type of stump: defective or not
* Type of amputation
* Circumstance of amputation: programmed / not programmed
* Psychological experience: Montgomery and Asberg Depression Scale score (MADRS)
* Socio-economic level
* The initial analgesic neuropathic treatment
* Possible previous prosthesis

It was also collected at week 4 and 8 :

- The level of advancement of the equipment by prosthesis

Each patient with the inclusion criteria, who agreed to participate in the study after reading the information note and signed consent, will be included in one of the two groups after randomization.

Group Reference Analgesic: receiving a reference antalgic management according to the protocol of the service: traditional management and treatment with Gabapentin.

Group Reference Analgesic and mirror therapy: receiving the reference antalgic management according to the protocol of the service: traditional management and treatment with Gabapentin as well as a management by mirror therapy during the first 4 weeks.

In group Reference analgesic and Mirror therapy, the mirror therapy will be performed by a physiotherapist trained in practice and already applying this technique in the center. Each patient receives, during the first week of treatment, 5 sessions of 20 minutes each decomposed as follows: 15 minutes of motor exercise and 5 minutes of sensory exercise. The content of the session was decided and put in place by the physiotherapist.

During the following 3 weeks the patients must practice self-rehabilitation at the rate of 5 sessions per week with a weekly re-evaluation session by the physiotherapist.

Before inclusion, the patient should be weaned as far as possible from neuropathic neuropathic treatments other than Gabapentin introduced for the treatment of phantom pain.

In both groups, patients receive the reference treatment according to the protocol of the service: titration of Gabapentin up to 3600 mg or maximum tolerated dose for 8 weeks.

Thereafter, depending on the patient's response and tolerance, the dose may be increased in increments of 300 mg / day every 2-3 days to a maximum dose of 3600 mg / day. A slower titration of gabapentin may be appropriate in some patients. The minimum time to reach a dose of 1800 mg / day is one week, to reach 2400 mg / day it is 2 weeks in total and to reach 3600 mg / day it is 3 weeks in total.

No other analgesic neuropathic treatment could be introduced or increased (PREGABALINE, AMITRIPTYLINE, DULOXETINE, MORPHINIC).

A punctual treatment (PARACETAMOL, CODEINE, NSAID, NEFOPAM) on acute pain without action on neuropathic type pain, linked to a different pathology is allowed.

If in Reference Analgesic group, the phantom limb pain was not sufficiently relieved at the end of the protocol, and the mirror therapy seems to be effective, a treatment by mirror therapy can be proposed to them.

The VAS and the details of the analgesic treatment will be collected every 2 weeks, blinded by an independent evaluator. Patients should not tell the evaluator which group they are assigned to.

The advancement of the prosthesis were collected at 4 and 8 weeks. Moreover, this is an observational study, following routine procedures already practiced systematically in the institution with this patient population. There are no additional procedures for diagnosis or additional medical supervision in this study.

16 subjects per group make it possible to demonstrate a size 1 effect with a risk of first species of 5% and a power of 80%. In order to take into account the risk of exiting the trial, we plan to include 20 patients in each group, sp a total of 40 patients.

Statistical analysis will use Sigma Plot® 12.5 for Windows Systat Software, Inc. or R software. Quantitative data will be reported in terms of mean, standard deviation and / or median and interquartile range. Qualitative data will be reported in terms of numbers and percentages.

The groups will be compared by Chi2 tests, or Fisher tests in case of insufficient numbers, for the qualitative variables. For quantitative variables the groups will be compared by T tests, or Wilcoxon tests if the variables do not have a normal distribution.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age who signed the memorandum.
* Patient hospitalized in the service for setting up equipment.
* In the aftermath of a major amputation of the lower limb, of vascular origin.
* Patients with phantom pain greater than or equal to 30 Visual Analog Evaluation (EVA); Whether pharmacologically or not.

Exclusion Criteria:

* Refusal to participate in the study.
* Presence of cognitive or psychiatric disorders that compromise the realization of mirror therapy.
* Presence of neurological, rheumatological or orthopedic disorders that may prevent movement of the unaffected limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the phantom limb pain using a VAS | 4 weeks
  The EVA and the details of the analgesic treatment were collected every two weeks, blinded by an independent evaluator. Patients should not tell the evaluator which group they are assigned to.

SECONDARY OUTCOMES:
Change from baseline of the Frequency of phantom limb pain episodes | every 2 weeks from day inclusion to Week 8
  Frequencies of painful attacks were collected every two weeks, blinded by an independent evaluator. Patients should not tell the evaluator which group they are assigned to.
change from baseline of the duration of phantom limb pain episodes. | every 2 weeks from day inclusion to Week 8
  Duration of painful attacks were collected every two weeks, blinded by an independent evaluator. Patients should not tell the evaluator which group they are assigned to.
Change from baseline of the consumption of pharmacological analgesic drugs | every 2 weeks from day inclusion to Week 8
  The consumption of pharmacological analgesic drugs were collected every two weeks, blinded by an independent evaluator. Patients should not tell the evaluator which group they are assigned to.
Quality of life? MEASUREMENT OF PAIN SENSATION | every 2 weeks from day inclusion to Week 8
  SF12
Sleep disorders | every 2 weeks from day inclusion to Week 8
  Spiegel Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Larlène Lacout, MD, Principal Investigator — APHP
Locations (1):
- Institut Merle d'Aubigné, Valenton, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] B Aledi L, Flumignan CD, Trevisani VF, Miranda F Jr. Interventions for motor rehabilitation in people with transtibial amputation due to peripheral arterial disease or diabetes. Cochrane Database Syst Rev. 2023 Jun 5;6(6):CD013711. doi: 10.1002/14651858.CD013711.pub2. PMID 37276273